CLINICAL TRIAL: NCT01647204
Title: Introduction of Mealtime Assistance Onto an Acute Medical Ward for Older People
Brief Title: Southampton Mealtime Assistance Study
Acronym: SMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09/H0502/93; RHM MED0882 (Other: UHS R&D ID)
Record Dates: First submitted 2012-07-11; First posted 2012-07-23 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Malnutrition
Keywords: Nutrition; older; hospital; volunteer
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual mealtime care (No Intervention): patients admitted to the control ward receiving no intervention but usual mealtime help from ward staff
- mealtime assistance (Experimental): Additional lunchtime help from trained volunteer mealtime assistants to supplement help from the ward staff
  Interventions: Other: trained volunteer mealtime assistance

INTERVENTIONS:
Other: trained volunteer mealtime assistance — trained volunteers helped inpatients at lunchtimes with dinner tray preparation, encouragement and feeding if required
  Arms: mealtime assistance

SUMMARY:
The primary objective of the study is to determine if the use of volunteers employed specifically to focus on mealtime assistance can increase food and nutrient intake of patients admitted to an acute Care of the Elderly ward. The sustainability of providing helpers to increase dietary intake over a year will be assessed and linked to actual dietary intake. The secondary objectives are to assess the association between dietary intake resulting from mealtime assistance and patient satisfaction, malnutrition risk, body composition, grip strength, length of hospital stay and hospital mortality.

DETAILED DESCRIPTION:
Poor nutritional status in older people acutely admitted to hospital is common with the risk of malnutrition estimated to be greater than 40%. Malnutrition is associated with major adverse clinical outcomes such as increased mortality, morbidity and length of stay at enormous cost to individuals and the health service. There is growing recognition that malnutrition is often unrecognised and untreated, and that many patients are discharged from hospital in a more malnourished state than when they were admitted. It is not surprising that complaints about nutrition and food services are amongst the commonest complaints in NHS hospitals.

The standard of mealtime care in UK hospitals has been an issue of concern for a number of years. A report last year from the Healthcare Commission found that one in five patients who wanted help eating did not get it. A secondary analysis of data provided by the Health Care Commission suggests that in some hospitals two out of five patients who wanted help with eating did not get it. Consistent with this, the recent Hungry to be Heard report found that nine out of ten nurses indicated they did not always have time to help ensure patients ate properly. They also suggested that some patients were not given appropriate assistance to eat. This problem is not unique to the UK and has been reported in other countries such as Australia and the USA.

The aim of the present study is to investigate if the use of volunteers employed specifically to focus on mealtime assistance in a Care of the Elderly Ward can increase food and nutrient intake, impact on body composition and improve clinical outcomes. The findings will inform service development in the nutritional care of older people across the Trust and wider.

ELIGIBILITY:
Inclusion Criteria:

Patients will be recruited in a consecutive prospective manner.

* emergency admissions to acute medical wards and
* ability to gain consent from patient or relatives

Exclusion Criteria:

* Patient acutely unwell or palliative care
* Patient lacking capacity to consent and no assent given by relatives
* Patients who are tube fed or nil-by-mouth

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 342 (Actual)
Dates: Start 2009-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
mean dietary intake of inpatients during a 24 hour period | end of year 1 and year 2
  The primary objective of the study is to determine if the use of volunteers employed specifically to focus on mealtime assistance can increase food and nutrient intake of patients admitted to an acute Care of the Elderly ward.
  Dietary intake measured as energy and protein

SECONDARY OUTCOMES:
patient satisfaction | end of year 1 and year2
  measured by patient interviews held during each year
malnutrition risk | end of year 1 and year2
  MUST score will be abstracted from medical records
length of stay in hospital | end of year one and year two
  taken from hospital records
grip strength | end of year 1 and year 2
  measured using a dynamometer
body composition | end of year one and year two and year 3
  triceps and mid upper arm measurement
mortality | end of year 1 year 2 and year 3
  abstracted from hospital records

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Roberts, MB ChB, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Roberts HC, Pilgrim AL, Jameson KA, Cooper C, Sayer AA, Robinson S. The Impact of Trained Volunteer Mealtime Assistants on the Dietary Intake of Older Female In-Patients: The Southampton Mealtime Assistance Study. J Nutr Health Aging. 2017;21(3):320-328. doi: 10.1007/s12603-016-0791-1. PMID 28244573
- [Derived] Roberts HC, Pilgrim AL, Elia M, Jackson AA, Cooper C, Sayer AA, Robinson SM. Southampton Mealtime Assistance Study: design and methods. BMC Geriatr. 2013 Jan 7;13:5. doi: 10.1186/1471-2318-13-5. PMID 23294981